CLINICAL TRIAL: NCT05073848
Title: Relationships Between Physical Activity and Different Measures of Fatigue in Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-3391.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-07-22; First posted 2021-10-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer Remission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BfitBwell Participants: Individuals in the BfitBwell Cancer Exercise Program complete a FACIT-Fatigue questionnaire at their baseline assessment. This will be screened for all incoming BfitBwell participants and those meeting the inclusion criteria of a score of 48 or less will be approached for interest in participating. The primary research activities beyond recruitment, screening, and informed consent are the collection of EMA fatigue assessments via smartphone application and PA assessment via actigraphy.

SUMMARY:
This is an investigation of possible relationships between daily physical activity (PA) and different measurements of fatigue in cancer survivors participating in a cancer exercise program.

DETAILED DESCRIPTION:
This is an investigation of possible relationships between daily physical activity (PA) and different measurements of fatigue in cancer survivors participating in a cancer exercise program. Results will inform exercise prescription and timing to best reduce fatigue, as well as methodology for measuring fatigue. Participants will answer several daily questions on fatigue using a smartphone application during the 3 month exercise program and wear a PA monitor for 10 days during the first month and last month of the program.

ELIGIBILITY:
Inclusion Criteria:

* Be an active participant in the BfitBwell Cancer Exercise Program
* Criteria for this program include:
* Adult (>= 18 years old)
* Being a patient seen at the University of Colorado Cancer Center
* Currently receiving cancer therapy or be within 6 months of completing cancer therapy
* Have a signed physician clearance form to participate in an exercise program
* Have a smartphone (necessary for the EMA assessments)
* A score of 48 or less on the FACIT-Fatigue (completed during the initial BfitBwell Program assessment)
* The minimally important difference of the FACIT-Fatigue is 3 points, suggesting that a score of at most 48 indicates the presence of CRF and allows for meaningful change in both directions.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 50-150 cancer survivors participating in the BfitBwell Cancer Exercise Program. As this is a non-invasive, exploratory observational investigation, there are minimal inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
10-point Fatigue Scale, Day | 3 months
  Severity of fatigue experienced over the course of the day, ranked 0-10. How would you rate your fatigue, over the last day, on a scale of 0-10, with 0 being no fatigue and 10 being the worst possible fatigue?
Physical Activity measure by Actigraph device | 3 months
  PA will be monitored using commonly used, non-invasive Actigraph devices (Actigraph GT3XP). Data will be collected utilizing methodology similar to that of the National Health and Nutrition Examination Survey (NHANES), in cancer survivors. The collected accelerometry data will be downloaded and analyzed in ActiLife software, calculation the average time spent in moderate-to-vigorous (MVPA) at each assessment period using standard algorithms and cut-points.

SECONDARY OUTCOMES:
Physical assessment measures from BfitBwell Program | 3 months
  As all participants are recruited from active members of BfitBwell Cancer Exercise Program, additional data will be extracted from program documents which are regularly administered and collected by the BfitBwell Program. Administration/collection will not change for study participants. Physical assessment measures are obtained from a physical assessment and electronic questionnaire.

OTHER OUTCOMES:
Response Rate to EMA assessments | 3 months
  Measures of fatigue are collected electronically. Tools utilized to collect these outcomes: REDCap and the LifeData smartphone application.
  * REDCap: REDCap is a secure, university supported and approved data collection tool. Links to complete the standardized questionnaires of fatigue (FACIT-Fatigue and MFI) will be emailed to participants with regular reminder emails sent daily until completed.
  * LifeData: LifeData is a secure research platform used by previous research studies involving EMA (https://www.lifedatacorp.com/customer-publications/). The application will send a smartphone notification to collect data at random timepoints in predefined windows, and allow participants to self-initiate data entry. Participants will not enter any identifying information and will instead be assigned a de-identified research IDd. Linking documentation of participant to this ID will be stored solely on university servers. LifeData will be utilized to collect the EMA assessments of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Marker, PhD, PT, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No